CLINICAL TRIAL: NCT00737243
Title: A Phase II Study of Chemotherapy Treatment Based on Molecular Profiling Diagnosis for Patients With Carcinoma of Unknown Primary Site
Brief Title: Treatment Based on Molecular Profiling Diagnosis Carcinoma of Unknown Primary Site
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI UNKPRI 20
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma
Keywords: Carcinoma of Unknown Primary Site; Molecular profiling assay; Bevacizumab; Erlotinib; Paclitaxel; Carboplatin
MeSH Terms: conditions — Carcinoma | interventions — Paclitaxel; Carboplatin; Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel, Carboplatin, Bevacizumab and Erlotinib (Experimental): Paclitaxel, Carboplatin, Bevacizumab and Erlotinib
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Bevacizumab; Drug: Erlotinib
- Treatment determined by physician (Other): Other treatment determined by physician based on molecular profiling assay
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Other: Treatment determined by physician

INTERVENTIONS:
Drug: Paclitaxel — 175 mg/m2, 1-3 hour IV infusion Day 1
  Arms: Paclitaxel, Carboplatin, Bevacizumab and Erlotinib
Drug: Carboplatin — AUC 6.0 IV Day 1
  Arms: Paclitaxel, Carboplatin, Bevacizumab and Erlotinib
Drug: Bevacizumab — 15 mg/kg IV infusion Day 1
  Other Names: Avastin
Drug: Erlotinib — 150 mg PO
  Other Names: Tarceva
Other: Treatment determined by physician — Patients Assigned a Specific Diagnosis by the Molecular profiling Assay will have physician's choice therapy
  Arms: Treatment determined by physician

SUMMARY:
This is a non-randomized Phase II study. Patients determined at initial diagnosis to have a carcinoma of unknown primary site (CUP) will have their treatment selected with the use of a molecular profiling assay. The assay will be performed on paraffin-embedded tumor tissue from a biopsy specimen. Patients given specific diagnoses (e.g., lung, pancreas, colon, breast, renal cell, prostate and ovarian cancer) will receive treatment regimens of proven activity. If no specific diagnosis is made with the molecular profiling assay, empiric chemotherapy with paclitaxel, carboplatin, bevacizumab and erlotinib will be administered.

DETAILED DESCRIPTION:
The primary objective of the study is evaluate the impact of the molecular assay prediction on the efficacy of therapy for patients with carcinoma of unknown primary site (CUP). Investigators will use tumor profiling results to direct standard, site-specific first-line therapy for patients with CUP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have carcinoma of unknown primary site after the following diagnostic procedures have been performed and are unrevealing of a primary site:

   * Complete medical history and physical examination,
   * Complete blood counts, chemistry profile,
   * CT scans of the chest and abdomen,
   * Directed evaluation of any symptomatic areas,
   * PET scan (recommended).
2. Patients must have biopsy-proven metastatic carcinoma, with any of the following light microscopic histologies:

   * Adenocarcinoma,
   * Poorly differentiated adenocarcinoma,
   * Poorly differentiated carcinoma (all patients with poorly differentiated carcinoma must have immunoperoxidase stains to rule out other treatable malignancies [e.g., lymphoma, neuroendocrine carcinoma]),
   * Poorly differentiated squamous carcinoma.
3. Patients must have biopsy material available from a surgical biopsy, a core needle biopsy, or a fine needle aspiration biopsy to provide an adequate specimen (must be 40% tumor) for the molecular profiling assay.
4. An ECOG performance status 0, 1, or 2.
5. No previous treatment with any systemic therapy.
6. Measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST).
7. Laboratory values as follows:

   * WBC 4000/micro L,
   * Platelets 100,000/micro L,
   * Serum bilirubin <1.5 times the institutional upper limits of normal (ULN),
   * Serum creatinine < 2.0 mg/dL.
8. Patients with brain metastases are eligible only if all lesions have been controlled by surgical resection or radiation therapy, the patient is not steroid-dependent, and the patient meets all other eligibility criteria.
9. Patients must be > 4 weeks from any major operative procedure.
10. To be eligible for the TREATMENT portion of the study, patients must have one of the five following diagnoses: colorectal, pancreas, NSCLC, ovary, renal cancer.
11. Patients must be able to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. Patients with the following specific syndromes are not eligible:

   * Patients with neuroendocrine carcinoma,
   * Women with adenocarcinoma isolated to axillary lymph nodes,
   * Women with adenocarcinoma isolated to peritoneal involvement,
   * Patients with carcinoma involving only 1 site, with resectable tumor at that site, or
   * Patients with squamous carcinoma limited to cervical, supraclavicular, or inguinal lymph nodes.
2. Patients with uncontrolled brain metastases and all patients with meningeal metastases.
3. Patients with insufficient biopsy material available for molecular profiling assay.
4. Women who are pregnant or lactating. All females of child-bearing potential must have a negative serum or urine pregnancy tests within 7 days prior to study treatment.
5. Men and women of childbearing potential are required to use effective methods of contraception during this study and for 6 months after ending therapy.
6. Patients who have received any other experimental drug within 28 days of starting treatment.

Exclusion Criteria for All Patients Receiving Bevacizumab-Containing Regimens

1. Patients with history of acute myocardial infarction within 6 months, other clinically significant cardiovascular disease (e.g., unstable angina, New York Heart Association [NYHA] grade 2 congestive heart failure [CHF], serious cardiac arrhythmias requiring medication) or > grade 2 vascular disease.
2. Patients with uncontrolled hypertension (systolic blood pressure [BP] 150 or diastolic BP >100mm Hg) or uncontrolled cardiac arrhythmias.
3. Prior hypertensive crisis or hypertensive encephalopathy.
4. Patients with clinical history of hemoptysis (defined as bright red blood of

   ½ teaspoon per episode) or hematemesis within 1 month prior to Day 1.
5. Patients with PEG tubes or G tubes.
6. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study.
7. Core biopsy or other minor surgical procedure excluding placement of a vascular access device, within 7 days prior to Day 1.
8. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1.
9. Patients with proteinuria (1000 mg/24 hours) at screening will be excluded. A 24-hour urine collection is not required in all patients (e.g., patients whose treatment plans exclude bevacizumab); however, all patients receiving bevacizumab with 1+ proteinuria on dipstick urinalysis at study entry must have a subsequent 24-hour urine collection.
10. Patients with any non-healing wound, ulcer, or long bone fracture.
11. Patients with any history of a bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
12. Patients with a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to beginning bevacizumab.
13. Patients with a history of stroke or transient ischemic attach within 6 months prior to first bevacizumab dose.
14. Known hypersensitivity to any component of bevacizumab.
15. Patients with history of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of a novel regimen, or that might affect the results of this study or render the subject at high risk for treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2008-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (21):
- United States (21):
  - Oncology Specialties (Clearview Cancer Institute), Huntsville, Alabama
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Baptist Hospital East, Louisville, Kentucky
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Jackson Oncology Associates, Jackson, Mississippi
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Derived] Hainsworth JD, Rubin MS, Spigel DR, Boccia RV, Raby S, Quinn R, Greco FA. Molecular gene expression profiling to predict the tissue of origin and direct site-specific therapy in patients with carcinoma of unknown primary site: a prospective trial of the Sarah Cannon research institute. J Clin Oncol. 2013 Jan 10;31(2):217-23. doi: 10.1200/JCO.2012.43.3755. Epub 2012 Oct 1. PMID 23032625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2008 and December 2011, 289 subjects in the United States with CUP were enrolled and had a molecular assay of biopsy tissue. 252 (87%) subjects had a successful assay performed; 223 subjects were treated and 29 were withdrawn (16 no longer met eligibility criteria and 13 were removed because of patient decision).
Pre-assignment Details: 252 subjects had successful assays. 223 subjects were treated and 29 were withdrawn prior to treatment. 194 received assay-directed therapy; 29 received empiric CUP therapy. Patients receiving assay-directed therapy were divided into 2 groups: 1) more responsive tumour type; and 2) less responsive tumour type.
Groups:
- All Patients With a Successful Tumor Assays Performed: Subjects in this group had a successful molecular assay of biopsy tissue
Period: Overall Study
Arm/Group | All Patients With a Successful Tumor Assays Performed
Started | 289
Successful Assay Performed | 252
Insufficient Tissue for Assay, Withdrawn | 37
Treated | 223
Not Treated | 29 (16 pts no longer met eligibility criteria; 13 came off study due to physician or pt preference.)
Site Specific Therapy More Responsive | 115
Site Specific Therapy Less Responsive | 79
Empiric CUP Therapy | 29
Completed | 194
Not Completed | 95

BASELINE CHARACTERISTICS:
Population: 252 patients who had successful assays.
Groups:
- Patients With Tumor Assays Performed: Of 289 patients initially enrolled, 252 had successful assays performed. 37 patients had insufficient tissue for assay and came off study.
Arm/Group | Patients With Tumor Assays Performed
Number analyzed (Participants) | 252
Age, Continuous [Median (Full Range); unit: years] | 64 [26 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 116
Region of Enrollment [Number; unit: participants]
  United States | 252

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Defined as the elapsed time from the start of treatment to the date of death from any cause or lost to follow-up. Participants lost to follow up were censored as of the last date known to be alive.
Time Frame: every 6-8 weeks (2 cycles) until death from any cause or lost to follow up, projected 18 months
Population: Of 223 treated patients: 194 received assay-directed therapy; 29 received empiric CUP therapy. The 194 patients who received assay-directed therapy were separated into groups based on predicted responsiveness of the tumor type for further analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- More Treatment Responsive: Patients who received assay-directed therapy for tumor types with a predicted median survival ≥ 12 months.
- Less Treatment Responsive: Patients who received assay-directed therapy for tumors with a predicted median survival ≤ 12 months
Arm/Group | More Treatment Responsive | Less Treatment Responsive
Number analyzed (Participants) | 115 | 79
months | 13.43 [10.57 to 16.03] | 7.62 [6.04 to 15.11]

2. Secondary Outcome: Number of Participants With a Tissue of Origin Successfully Predicted by the Assay
Description: To evaluate the utility of the assay in identifying the tissue of origin in patients with carcinoma of unknown primary site (CUP), an archived tumor specimen was assayed upon study entry. If a tissue of origin was predicted by the assay, participants received standard site-specific therapy for that tumor type. When tissue of origin was not predicted by the assay, patients received standard empiric chemotherapy for CUP and were not followed further. If the assay was not completed due to inadequate amount of tumor in the biopsy specimen, patients were not treated on the study.
Time Frame: at baseline
Population: Of 252 participants analyzed, the assay correctly predicted the tissue of origin in 247 patients (98%). The predicted tissue of origin could not be determined in 5 participants (2%).
Measure: Number; unit: participants
Groups:
- Patients With Successful Tumor Assays Performed: In 252 participants successful assays were performed. In 29 participants the amount of tumour and/or viable RNA present in the biopsy specimen was inadequate.
Arm/Group | Patients With Successful Tumor Assays Performed
Number analyzed (Participants) | 252
participants
  Biliary tract (gallbladder, bile duct) | 52
  Urothelium | 31
  Colorectum | 28
  Non-small cell lung | 27
  Pancreas | 12
  Breast | 12
  Ovary | 11
  Gastroesophageal | 10
  Kidney | 9
  Liver | 8
  Sarcoma | 6
  Cervix | 6
  Neuroendocrine | 5
  Prostate | 4
  Germ cell | 4
  Skin, squamous | 4
  Carcinoid, intestine | 3
  Mesothelioma | 3
  Thyroid | 2
  Endometrium | 2
  Melanoma | 2
  Skin, basal-cell | 2
  Lung, small-cell | 1
  Lymphoma | 1
  Head and Neck | 1
  Adrenal | 1
  unclassifiable | 5

ADVERSE EVENTS:
Time Frame: every 6-8 weeks (2 cycles) up to 48 weeks
Description: Adverse event data were collected for 223 participants treated with at least one dose of study drug.
Arm/Group | All Treated Patients
Serious Adverse Events (participants affected / at risk) | 30/223
Other Adverse Events (participants affected / at risk) | 74/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Patients (N=223)
Abdominal pain (Gastrointestinal disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac disorders - Other, left ventricular diastolic dysfunction (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Esophageal ulcer (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 1
Gastrointestinal disorders - Other, small bowel obstruction (Gastrointestinal disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hepatobiliary disorders - Other, hepatic dysfunction (Hepatobiliary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, infection at port site (Infections and infestations) | 2
Infections and infestations - Other, pneumonia (Infections and infestations) | 1
Infections and infestations - Other, unspecified (Infections and infestations) | 1
INR increased (Investigations) | 1
Ischemia cerebrovascular (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Platelet count decreased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Thromboembolic event (Vascular disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Patients (N=223)
Platelet count decreased (Investigations) | 22
Fatigue (General disorders) | 21
Neutrophil count decreased (Investigations) | 18
Anemia (Blood and lymphatic system disorders) | 15
White blood cell decreased (Investigations) | 14

LIMITATIONS AND CAVEATS:
The focus of this study was to evaluate the ability of the 92-gene assay to successfully predict tumor tissue of origin, not to assess one particular treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites